CLINICAL TRIAL: NCT00605475
Title: A Multi Center, Randomized, Double Blind, Placebo-controlled, Dose Escalation Study of the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ACZ885 Administered Intravenously to Patients With Type 2 Diabetes Mellitus
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ACZ885 in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CACZ885A2213
Record Dates: First submitted 2008-01-18; First posted 2008-01-31 (Estimated); Results first posted 2012-02-13 (Estimated); Last update posted 2012-02-13 (Estimated); Status verified 2012-01

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus; Canakinumab; ACZ885; IL-1B antagonist; metformin; glycemic control; insulin sensitivity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — canakinumab; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Canakinumab (Experimental): Eligible participants were assigned to receive canakinumab in one of four cohorts; 1) Single IV infusion of canakinumab 0.3 mg/kg; 2) Singe IV infusion of canakinumab 10 mg/kg; 3) single IV infusion of canakinumab 0.1 mg/kg or 0.3 mg/kg, or 1.5 mg/kg; 4) Single IV injection of canakinumab 0.03 mg/kg.
  All participants were required to take a concomitant stable daily dose of metformin during the study.
  Interventions: Drug: Canakinumab; Drug: Metformin
- Placebo (Placebo Comparator): Eligible participants were assigned to receive placebo to canakinumab in one of four cohorts; 1) Single IV infusion of placebo to canakinumab 0.3 mg/kg; 2) Singe IV infusion of placebo to canakinumab 10 mg/kg; 3) single IV infusion of placebo to canakinumab 0.1 mg/kg or 0.3 mg/kg, or 1.5 mg/kg; 4) Single IV injection of placebo to canakinumab 0.03 mg/kg.
  All participants were required to take a concomitant stable daily dose of metformin during the study.
  Interventions: Drug: Placebo; Drug: Metformin

INTERVENTIONS:
Drug: Canakinumab — Canakinumab given as single dose IV injection of 0.03 mg/kg, or single dose IV infusion at doses of 0.1 mg/kg 0.3 mg/kg, 1.5 mg/kg or 10 mg/kg.
  Other Names: ACZ885
  Arms: Canakinumab
Drug: Placebo — Placebo to Canakinumab given as single dose IV injection of 0.03 mg/kg, or single dose IV infusion at doses of 0.1 mg/kg 0.3 mg/kg, 1.5 mg/kg or 10 mg/kg.
  Arms: Placebo
Drug: Metformin — Participants continued on their stable daily dose of metformin throughout the study
  Other Names: Glucophage; Glumetza

SUMMARY:
The purpose of this study was to evaluate, in patients with Type 2 Diabetes Mellitus, whether Canakinumab can lower Glycosylated hemoglobin / hemoglobin A1c (HbA1c) and/or peak glucose levels in response to an oral glucose tolerance test (OGTT).

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 18 to 70 years, with type 2 diabetes mellitus (non-insulin dependent diabetes) for at least 6 months prior to study start
* HbA1c between 7.0 and 9.5%
* On stable dose metformin monotherapy
* Stable body weight

Exclusion Criteria:

* Poorly controlled type 2 diabetes (very low or very high blood sugar levels, or other indicators of poor control)
* Acute infections prior to dosing
* Patients with type 1 diabetes (insulin-dependent diabetes)
* Taking diabetes medication (other than metformin)

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2007-12; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: NOVARTIS, Principal Investigator — Novartis investigator site
Locations (13):
- United States (6):
  - Arkansas Research Medical Testing, Little Rock, Arkansas
  - Allied Research International - Cetero Research Miami, Miami, Florida
  - Elite Research Institute Miami, Miami, Florida
  - International Research Center Towson, MD, Maryland
  - Covance Clinical Research Unit Inc, Portland, Oregon
  - Charles River Clinical Services, Northwest Tacoma, Washington
- Germany (5):
  - Novartis Investigator Site, Berlin
  - Novartis Investigator Site, Kiel
  - Novartis Investigator Site, Mönchengladbach
  - Novartis Investigator Site, Munich
  - Novartis Investigative Site, Neuss
- Russia (2):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersberg

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Canakinumab Infusion 0.3 mg/kg: Single dose intravenous (IV) infusion of canakinumab 0.3 mg/kg
- Cohort 1: Placebo to Canakinumab 0.3 mg/kg: Single dose IV infusion of placebo to Canakinumab 0.3 mg/kg
- Cohort 2: Canakinumab Infusion 10 mg/kg: Single dose IV infusion of Canakinumab 10 mg/kg
- Cohort 2: Placebo to Canakinumab 10 mg/kg: Single dose IV infusion of Placebo to Canakinumab 10 mg/kg
- Cohort 3: Canakinumab Infusion 0.1 mg/kg: Single dose IV infusion Canakinumab 0.1 mg/kg
- Cohort 3: Canakinumab Infusion 0.3 mg/kg: Single dose IV infusion of Canakinumab 0.3 mg/kg
- Cohort 3 : Canakinumab Infusion 1.5 mg/kg: Single dose IV infusion of canakinumab 1.5 mg/kg
- Cohort 3: Placebo Infusion: Single dose IV infusion of Placebo
- Cohort 4 : Canakinumab Injection 0.03 mg/kg: Single dose IV injection of Canakinumab 0.03 mg/kg
- Cohort 4: Placebo to Canakinumab 0.03 mg/kg: Single dose IV injection of Placebo to Canakinumab 0.03 mg/kg
Period: Overall Study
Arm/Group | Cohort 1: Canakinumab Infusion 0.3 mg/kg | Cohort 1: Placebo to Canakinumab 0.3 mg/kg | Cohort 2: Canakinumab Infusion 10 mg/kg | Cohort 2: Placebo to Canakinumab 10 mg/kg | Cohort 3: Canakinumab Infusion 0.1 mg/kg | Cohort 3: Canakinumab Infusion 0.3 mg/kg | Cohort 3 : Canakinumab Infusion 1.5 mg/kg | Cohort 3: Placebo Infusion | Cohort 4 : Canakinumab Injection 0.03 mg/kg | Cohort 4: Placebo to Canakinumab 0.03 mg/kg
Started | 10 | 5 | 45 | 45 | 25 | 24 | 23 | 24 | 20 | 10
Completed | 10 | 5 | 45 | 45 | 24 | 22 | 22 | 24 | 18 | 8
Not Completed | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 2 | 2
Not completed — Abnormal Laboratory Values | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Administrative problems | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Canakinumab Infusion 0.3 mg/kg | Cohort 1: Placebo to Canakinumab 0.3 mg/kg | Cohort 2: Canakinumab Infusion 10 mg/kg | Cohort 2: Placebo to Canakinumab 10 mg/kg | Cohort 3: Canakinumab Infusion 0.1 mg/kg | Cohort 3: Canakinumab Infusion 0.3 mg/kg | Cohort 3 : Canakinumab Infusion 1.5 mg/kg | Cohort 3: Placebo Infusion | Cohort 4 : Canakinumab Injection 0.03 mg/kg | Cohort 4: Placebo to Canakinumab 0.03 mg/kg | Total
Number analyzed (Participants) | 10 | 5 | 45 | 45 | 25 | 24 | 23 | 24 | 20 | 10 | 231
Age Continuous [Mean (Standard Deviation); unit: years] | 53 (7.60) | 52 (6.96) | 57.1 (9.38) | 57.5 (7.95) | 53.9 (7.58) | 55 (8.45) | 55.1 (9.28) | 54.7 (6.41) | 53.9 (9.07) | 56 (8.67) | 54.6 (8.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 21 | 14 | 13 | 17 | 14 | 16 | 10 | 2 | 116
  Male | 4 | 2 | 24 | 31 | 12 | 7 | 9 | 8 | 10 | 8 | 115

OUTCOME MEASURES:

1. Secondary Outcome: Mean Change From Baseline in Plasma C-peptide AUC ( Area Under the Curve) 0-4 Hours, Following Oral Glucose Tolerance Test (OGTT)
Description: Blood samples were drawn after an overnight fast and standard OGTT at 0, 15, 30, 45, 60, 90, 120, 180 and 240 min. C-peptide levels over 4 hrs were shown as Area Under the Curve, (AUC). Analysis of covariance with treatment as a fixed effect and baseline as the covariate was performed.
Time Frame: Baseline, Day 28, Day 84
Population: All randomized participants who received study drug were included in the intent to treat population (ITT). Last observation carried forward (LOCF) was used to impute missing values.
Measure: Least Squares Mean (Standard Error); unit: pmol*h/L
Groups:
- Cohort 2: Placebo to Canakinumab 10 mg/kg: Single dose IV infusion of Canakinumab 10 mg/kg
- Cohort 3: Canakinumab Infusion 1.5 mg/kg: Single dose IV infusion of canakinumab 1.5 mg/kg
- Pooled (Cohort 3 and 4): Placebo Infusion: Pooled Placebo of Cohort 3 and 4. Single dose IV infusion of Placebo
- Cohort 4: Canakinumab Injection 0.03 mg/kg: Single dose IV injection of Canakinumab 0.03 mg/kg
Arm/Group | Cohort 2: Canakinumab Infusion 10 mg/kg | Cohort 2: Placebo to Canakinumab 10 mg/kg | Cohort 3: Canakinumab Infusion 0.1 mg/kg | Cohort 3: Canakinumab Infusion 0.3 mg/kg | Cohort 3: Canakinumab Infusion 1.5 mg/kg | Pooled (Cohort 3 and 4): Placebo Infusion | Cohort 4: Canakinumab Injection 0.03 mg/kg
Number analyzed (Participants) | 45 | 45 | 25 | 24 | 23 | 34 | 20
pmol*h/L
  Day 28 (n= 41, 41, 21, 23, 23, 31, 20) | -335 (178.1) | -614 (178.1) | -492 (392.4) | -25 (367.6) | 779 (367.6) | 129 (319.4) | -553 (394.6)
  Day 84 (n= 41, 43, 22, 24, 23, 32, 20) | -601 (275.1) | -205 (268.6) | 143 (386.5) | 143 (361.1) | 654 (368.9) | 240 (316.0) | -939 (396.1)

2. Primary Outcome: Mean Change From Baseline in Plasma HbA1c (Glycosylated Hemoglobin / Hemoglobin A1c)
Description: Blood was drawn after an overnight fast to measure plasma HbA1c levels. End of Study is defined as the last Analysis of covariance with treatment as a fixed effect and baseline as the covariate was performed.
Time Frame: Baseline, Day 28, Day 84, Day 126, End of Study (168 [+/- 5] days after dosing)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent
Groups:
- Cohort 2:Placebo to Canakinumab 10 mg/kg: Single dose IV infusion of Canakinumab 10 mg/kg
Arm/Group | Cohort 2: Canakinumab Infusion 10 mg/kg | Cohort 2:Placebo to Canakinumab 10 mg/kg | Cohort 3: Canakinumab Infusion 0.1 mg/kg | Cohort 3: Canakinumab Infusion 0.3 mg/kg | Cohort 3: Canakinumab Infusion 1.5 mg/kg | Pooled (Cohort 3 and 4): Placebo Infusion | Cohort 4: Canakinumab Injection 0.03 mg/kg
Number analyzed (Participants) | 45 | 45 | 25 | 24 | 23 | 34 | 20
percent
  Day 28 (n= 45, 45, 25, 23, 23, 34, 20) | -0.38 (0.057) | -0.26 (0.057) | -0.25 (0.065) | -0.30 (0.069) | -0.47 (0.068) | -0.24 (0.056) | -0.13 (0.073)
  Day 84 (n= 44, 44, 25, 23, 23, 33, 20) | -0.46 (0.102) | -0.15 (0.105) | -0.04 (0.118) | -0.43 (0.124) | -0.59 (0.124) | 0.32 (0.103) | -0.15 (0.132)
  Day 126 (n= 45, 45, 21, 22, 23, 33, 20) | -0.29 (0.101) | -0.02 (0.101) | -0.08 (0.126) | -0.22 (0.123) | -0.40 (0.120) | -0.19 (0.101) | -0.11 (0.128)
  End of Study (n= 43, 45, 24, 20, 21, 33, 20) | -0.26 (0.121) | -0.01 (0.118) | 0.27 (0.162) | -0.18 (0.178) | -0.39 (0.173) | -0.12 (0.138) | 0.32 (0.177)

3. Secondary Outcome: Mean Change From Baseline in Plasma Insulin AUC ( Area Under the Curve) 0-4 Hours, Following Oral Glucose Tolerance Test ( OGTT )
Description: Blood samples were drawn after an overnight fast and OGTT at 0, 15, 30, 45, 60, 90, 120, 180 and 240 min. Insulin levels over 4 hrs were shown as Area Under the Curve, (AUC). Analysis of covariance with treatment as a fixed effect and baseline as the covariate was performed.
Time Frame: Baseline, Day 28, Day 84
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: µIU*h/mL
Groups:
- Pooled (Cohort 3 and 4): Placebo Infusion: Pooled placebo from Cohort 3 and 4. Single dose IV infusion of Placebo
Arm/Group | Cohort 2: Canakinumab Infusion 10 mg/kg | Cohort 2: Placebo to Canakinumab 10 mg/kg | Cohort 3: Canakinumab Infusion 0.1 mg/kg | Cohort 3: Canakinumab Infusion 0.3 mg/kg | Cohort 3: Canakinumab Infusion 1.5 mg/kg | Pooled (Cohort 3 and 4): Placebo Infusion | Cohort 4: Canakinumab Injection 0.03 mg/kg
Number analyzed (Participants) | 45 | 45 | 25 | 24 | 23 | 34 | 20
µIU*h/mL
  Day 28 (n= 43, 45, 18, 21,16, 29, 20) | -1.58 (6.156) | -14.25 (6.017) | -12.61 (8.173) | 6.06 (7.477) | 2.06 (8.494) | -8.26 (6.421) | -1.35 (7.637)
  Day 84 (n= 43, 45, 22, 23, 19, 31, 20) | -19.68 (11.054) | -6.97 (10.805) | -8.38 (9.095) | 2.44 (8.673) | -6.65 (9.522) | -4.09 (7.592) | -10.52 (9.321)

4. Secondary Outcome: Mean Change From Baseline in Plasma Proinsulin AUC ( Area Under the Curve) 0-4 Hours, Following Oral Glucose Tolerance Test ( OGTT )
Description: as for outcome 3
Time Frame: Baseline, Day 28, Day 84
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: pmol*h/L
Groups:
- Pooled (Cohort 3 and 4): Placebo Infusion: Pooled placebo from cohort 3 and 4. ingle dose IV infusion of Placebo
Arm/Group | Cohort 2: Canakinumab Infusion 10 mg/kg | Cohort 2: Placebo to Canakinumab 10 mg/kg | Cohort 3: Canakinumab Infusion 0.1 mg/kg | Cohort 3: Canakinumab Infusion 0.3 mg/kg | Cohort 3: Canakinumab Infusion 1.5 mg/kg | Pooled (Cohort 3 and 4): Placebo Infusion | Cohort 4: Canakinumab Injection 0.03 mg/kg
Number analyzed (Participants) | 45 | 45 | 25 | 24 | 23 | 34 | 20
pmol*h/L
  Day 28 (n= 36, 37, 22, 24, 21, 30, 20) | -9.9 (8.37) | 11.0 (8.25) | -13.7 (18.78) | -15.0 (17.64) | 26.1 (18.81) | -16.2 (16.38) | -22.3 (19.25)
  Day 84 (n= 36, 37, 23, 24, 21, 30, 20) | -6.2 (10.95) | 7.8 (10.79) | -25.8 (20.96) | -9.3 (20.33) | 39.6 (21.68) | -25.9 (18.76) | -17.3 (22.17)

5. Secondary Outcome: Mean Change From Baseline in Plasma Glucagon AUC ( Area Under the Curve) 0-4 Hours, Following Oral Glucose Tolerance Test
Description: Blood samples were drawn after an overnight fast and OGTT at 0, 15, 30, 45, 60, 90, 120, 180 and 240 min. Glucagon levels over 4 hrs were shown as Area Under the Curve, (AUC). Analysis of covariance with treatment as a fixed effect and baseline as the covariate was performed.
Time Frame: Baseline, Day 28, Day 84
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: pmol*h/L
Groups:
- Pooled (Cohort 3 and 4) Placebo Infusion: Pooled placebo from cohort 3 and 4. Single dose IV infusion of Placebo
Arm/Group | Cohort 2: Canakinumab Infusion 10 mg/kg | Cohort 2: Placebo to Canakinumab 10 mg/kg | Cohort 3: Canakinumab Infusion 0.1 mg/kg | Cohort 3: Canakinumab Infusion 0.3 mg/kg | Cohort 3: Canakinumab Infusion 1.5 mg/kg | Pooled (Cohort 3 and 4) Placebo Infusion | Cohort 4: Canakinumab Injection 0.03 mg/kg
Number analyzed (Participants) | 45 | 45 | 25 | 24 | 23 | 34 | 20
pmol*h/L
  Day 28 (n= 41, 44, 22, 23, 23, 34, 20) | -3.6 (2.30) | -4.0 (2.22) | -3.1 (3.43) | -3.7 (3.37) | -0.6 (3.36) | -2.7 (2.78) | -5.5 (3.60)
  Day 84 (n= 42, 45, 23, 23, 23, 33, 20) | -3.7 (2.96) | -2.0 (2.86) | -1.0 (4.46) | -1.8 (4.48) | 14.7 (4.46) | 2.9 (3.74) | -4.0 (4.79)

6. Primary Outcome: Mean Change From Baseline in Plasma Glucose Area Under the Curve (AUC) 0 - 4 Hours Following Oral Glucose Tolerance Test (OGTT )
Description: Mean Change in Glucose level stimulated by OGTT. Blood samples were taken at sample times: -20, -10, -1 and 10, 20, 30, 60, 90, 120, 180, and 240 minutes. Glucose levels over 4 hrs were shown as Area Under the Curve, (AUC). Analysis of covariance with treatment as a fixed effect and baseline as the covariate was performed.
Time Frame: Baseline, Day 28, Day 84
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol*h/L
Groups:
- Pooled (Cohort 3and 4): Placebo Infusion: Pooled Placebo of Cohort 3 and 4. Single dose IV infusion of Placebo
Arm/Group | Cohort 2: Canakinumab Infusion 10 mg/kg | Cohort 2: Placebo to Canakinumab 10 mg/kg | Cohort 3: Canakinumab Infusion 0.1 mg/kg | Cohort 3: Canakinumab Infusion 0.3 mg/kg | Cohort 3: Canakinumab Infusion 1.5 mg/kg | Pooled (Cohort 3and 4): Placebo Infusion | Cohort 4: Canakinumab Injection 0.03 mg/kg
Number analyzed (Participants) | 43 | 45 | 24 | 24 | 22 | 33 | 20
mmol*h/L
  Day 28 | -4.7 (0.98) | -0.9 (0.96) | 1.6 (1.66) | -0.9 (1.65) | -2.8 (1.73) | -2.3 (1.41) | -0.5 (1.81)
  Day 84 | -2.5 (1.26) | 1.7 (1.24) | 2.6 (1.72) | -2.8 (1.71) | -1.2 (1.79) | -2.8 (1.46) | -2.5 (1.88)

7. Secondary Outcome: Mean Change From Baseline in Peak Plasma Insulin/Proinsulin Level, Following Oral Glucose Tolerance Test (OGTT)
Description: Blood samples were drawn after an overnight fast and OGTT at 0, 15, 30, 45, 60, 90, 120, 180 and 240 min. Insulin and proinsulin levels were measured. The insulin/proinsulin level was calculated by dividing the insulin level by the proinsulin level. Analysis of covariance with treatment as a fixed effect and baseline as the covariate was performed.
Time Frame: Baseline, Day 28, Day 84
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: pmol/pmol
Groups:
- Cohort 4:Canakinumab Injection 0.03 mg/kg: Single dose IV injection of Canakinumab 0.03 mg/kg
Arm/Group | Cohort 2: Canakinumab Infusion 10 mg/kg | Cohort 2: Placebo to Canakinumab 10 mg/kg | Cohort 3: Canakinumab Infusion 0.1 mg/kg | Cohort 3: Canakinumab Infusion 0.3 mg/kg | Cohort 3: Canakinumab Infusion 1.5 mg/kg | Pooled (Cohort 3 and 4): Placebo Infusion | Cohort 4:Canakinumab Injection 0.03 mg/kg
Number analyzed (Participants) | 45 | 45 | 25 | 24 | 23 | 34 | 20
pmol/pmol
  Day 28 (n= 43, 45, 24, 24, 23, 34,20) | 0.173 (0.3902) | -1.035 (0.3814) | 0.160 (0.7996) | 1.039 (0.7996) | 0.293 (0.8169) | -0.031 (0.6755) | 0.518 (0.8832)
  Day 84 (n= 44, 44, 25, 24, 23, 34, 20) | -0.852 (0.4890) | -0.688 (0.4890) | -0.689 (0.7973) | 0.923 (0.8138) | 0.250 (0.8313) | 0.682 (0.6871) | -0.046 (0.8991)

8. Secondary Outcome: Mean Insulin Secretion Rate ( ISR ) Relative to Glucose, 0 - 4 Hours
Description: Blood samples were taken at sample times: -20, -10, -1 and 10, 20, 30, 60, 90, 120, 180, and 240 minutes. Mean ISR relative to glucose over 0-4 hours was calculated as follows:
  Mean ISR relative to glucose = mean ISR / (glucose AUC/time interval). The mean ISR was computed as an AUC (area under the curve) using the linear trapezoidal rule divided by the corresponding time interval. Analysis of covariance with treatment as a fixed effect and baseline as the covariate was performed.
Time Frame: Day 28, Day 84
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: pmol/min/m^2/mmol/L
Groups:
- Canakinumab Injection 0.03 mg/kg: Single dose IV injection of Canakinumab 0.03 mg/kg
Arm/Group | Cohort 2: Canakinumab Infusion 10 mg/kg | Cohort 2: Placebo to Canakinumab 10 mg/kg | Cohort 3: Canakinumab Infusion 0.1 mg/kg | Cohort 3: Canakinumab Infusion 0.3 mg/kg | Cohort 3: Canakinumab Infusion 1.5 mg/kg | Pooled (Cohort 3 and 4) Placebo Infusion | Canakinumab Injection 0.03 mg/kg
Number analyzed (Participants) | 45 | 45 | 25 | 24 | 23 | 34 | 20
pmol/min/m^2/mmol/L
  Day 28 (n= 41, 43, 23, 23, 22, 33, 20) | 20.4 (0.53) | 18.0 (0.52) | 14.5 (1.03) | 17.1 (1.03) | 19.1 (1.05) | 18.5 (0.86) | 16.1 (1.10)
  Day 84 (n= 42, 43, 24, 24, 22, 33, 20) | 18.5 (1.00) | 19.0 (0.99) | 16.8 (1.13) | 18.4 (1.13) | 18.5 (1.18) | 18.9 (0.96) | 15.9 (1.24)

9. Secondary Outcome: Mean Insulin Secretion Rate ( ISR ), 0 - 4 Hours
Description: Blood samples were taken at sample times: -20, -10, -1 and 10, 20, 30, 60, 90, 120, 180, and 240 minutes. The mean ISR over 0 - 4 hours was computed as an AUC (area under the curve) using the linear trapezoidal rule divided by the corresponding time interval. Analysis of covariance with treatment as a fixed effect and baseline as the covariate was performed.
Time Frame: Day 28, Day 84
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: pmol/min/m^2
Arm/Group | Cohort 2: Canakinumab Infusion 10 mg/kg | Cohort 2: Placebo to Canakinumab 10 mg/kg | Cohort 3: Canakinumab Infusion 0.1 mg/kg | Cohort 3: Canakinumab Infusion 0.3 mg/kg | Cohort 3: Canakinumab Infusion 1.5 mg/kg | Pooled (Cohort 3 and 4) Placebo Infusion | Canakinumab Injection 0.03 mg/kg
Number analyzed (Participants) | 45 | 45 | 25 | 24 | 23 | 34 | 20
pmol/min/m^2
  Day 28 (n= 42, 43, 23, 23, 23, 33, 20) | 255 (6.4) | 246 (6.3) | 207 (13.1) | 231 (13.0) | 262 (13.0) | 234 (10.9) | 212 (13.9)
  Day 84 (n= 43, 43, 25, 24, 23, 34, 20) | 248 (9.3) | 259 (9.3) | 234 (12.6) | 234 (12.7) | 254 (13.0) | 239 (10.8) | 197 (13.9)

10. Secondary Outcome: Insulin Sensitivity Index ( ISI ) at Day 28, Day 48
Description: Insulin sensitivity index (ISI) = 10000 / [fasting insulin (μIU/mL) x fasting glucose (mg/dL) x mean 2 hour insulin(μIU/mL) x mean 2 hour glucose (mg/dL)]1/2 where mean 2 hour insulin (or glucose) was defined as the insulin (or glucose)AUC(0-2 hr) divided by the time period (2 hr). In normal subjects the mean score ± SE is 0.366 ± 0.029. Analysis of covariance with treatment as a fixed effect and baseline as the covariate was performed on log transformed data.
Time Frame: Day 28, Day 84
Population: as for outcome 1
Measure: Geometric Mean (Standard Error); unit: units on a scale
Arm/Group | Cohort 2: Canakinumab Infusion 10 mg/kg | Cohort 2: Placebo to Canakinumab 10 mg/kg | Cohort 3: Canakinumab Infusion 0.1 mg/kg | Cohort 3: Canakinumab Infusion 0.3 mg/kg | Cohort 3: Canakinumab Infusion 1.5 mg/kg | Pooled (Cohort 3 and 4): Placebo Infusion | Cohort 4: Canakinumab Injection 0.03 mg/kg
Number analyzed (Participants) | 45 | 45 | 25 | 24 | 23 | 34 | 20
units on a scale
  Day 28 (n= 40, 40, 12, 17, 14, 22, 20) | 2.91 (0.049) | 2.63 (0.049) | 3.13 (0.093) | 2.96 (0.077) | 3.57 (0.083) | 3.77 (0.068) | 3.39 (0.071)
  Day 84 (n= 39, 43, 13, 20, 14, 27, 20) | 2.96 (0.043) | 2.80 (0.041) | 3.34 (0.109) | 3.04 (0.085) | 2.99 (0.101) | 3.63 (0.074) | 3.70 (0.086)

11. Secondary Outcome: Insulinogenic Index, 0 - 30 Minutes
Description: Insulinogenic index (0-30 min)
  * [Change in insulin (0-30 min) (μIU/mL)] / [Change in glucose (0-30 min) (mg/dL)]
  * [insulin (μIU/mL) at 30 min - insulin (μIU/mL) at 0 min] / [glucose (mg/dL) at 30 min - glucose (mg/dL) at 0 min), where insulin (or glucose) at 0 min was defined as the arithmetic mean of the -15, -10 and 0 min pre-glucose load values. Analysis of covariance with treatment as a fixed effect and baseline as the covariate was performed on log transformed data..
Time Frame: Day 28, Day 84
Population: as for outcome 1
Measure: Geometric Mean (Standard Error); unit: units on a scale
Arm/Group | Cohort 2: Canakinumab Infusion 10 mg/kg | Cohort 2: Placebo to Canakinumab 10 mg/kg | Cohort 3: Canakinumab Infusion 0.1 mg/kg | Cohort 3: Canakinumab Infusion 0.3 mg/kg | Cohort 3: Canakinumab Infusion 1.5 mg/kg | Pooled (Cohort 3 and 4): Placebo Infusion | Cohort 4: Canakinumab Injection 0.03 mg/kg
Number analyzed (Participants) | 45 | 45 | 25 | 24 | 23 | 34 | 20
units on a scale
  Day 28 (n=44, 44, 17, 23 17, 32, 18) | 0.174 (0.0754) | 0.140 (0.0754) | 0.090 (0.1995) | 0.105 (0.1735) | 0.139 (0.1991) | 0.102 (0.1464) | 0.137 (0.1942)
  Day 84 (n=43, 44, 17, 24, 20, 31, 17) | 0.157 (0.0987) | 0.134 (0.0976) | 0.092 (0.1928) | 0.098 (0.1651) | 0.111 (0.1777) | 0.124 (0.1445) | 0.121 (0.1937)

12. Secondary Outcome: Mean Change From Baseline in Peak Plasma Glucose Following Oral Glucose Tolerance Test ( OGTT )
Description: Mean Change in Peak Glucose level stimulated by OGTT. Blood samples were taken at sample times: -20, -10, -1 and 10, 20, 30, 60, 90, 120, 180, and 240 minutes. Change from baseline assessed at Day 28 and 84. Analysis of covariance with treatment as a fixed effect and baseline as the covariate was performed.
Time Frame: Baseline, Day 28, Day 84
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Groups:
- Cohort 3:Canakinumab Infusion 0.3 mg/kg: Single dose IV infusion of Canakinumab 0.3 mg/kg
- Cohort 3:Canakinumab Infusion 1.5 mg/kg: Single dose IV infusion of canakinumab 1.5 mg/kg
Arm/Group | Cohort 2: Canakinumab Infusion 10 mg/kg | Cohort 2: Placebo to Canakinumab 10 mg/kg | Cohort 3: Canakinumab Infusion 0.1 mg/kg | Cohort 3:Canakinumab Infusion 0.3 mg/kg | Cohort 3:Canakinumab Infusion 1.5 mg/kg | Pooled (Cohort 3 and 4) Placebo Infusion | Cohort 4:Canakinumab Injection 0.03 mg/kg
Number analyzed (Participants) | 44 | 45 | 24 | 24 | 23 | 33 | 20
mmol/L
  Day 28 | -1.3 (0.30) | 0.0 (0.30) | 0.2 (0.55) | -0.2 (0.55) | -0.8 (0.57) | -1.0 (0.47) | 0.1 (0.61)
  Day 84 | -0.9 (0.38) | 0.6 (0.37) | 0.2 (0.58) | -0.7 (0.58) | 0.3 (0.60) | -0.9 (0.50) | -0.3 (0.64)

13. Secondary Outcome: Mean Change From Baseline in Peak Plasma Fructosamine Level
Description: Blood was drawn to measure change in plasma Fructosamine Level, from baseline to Day 14, 28, 56, 84, 126 and End of Study ( defined as the final available post-randomization assessment up to the last regularly scheduled visit at Day 168 [+/- 5]). Analysis of covariance with treatment as a fixed effect and baseline as the covariate was performed.
Time Frame: Baseline, Day 14, Day 28, Day 56, Day 84, Day 126, End of Study (168 [+/- 5] days after dosing)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: µmol/L
Arm/Group | Cohort 2: Canakinumab Infusion 10 mg/kg | Cohort 2: Placebo to Canakinumab 10 mg/kg
Number analyzed (Participants) | 45 | 45
µmol/L
  Day 14 (n= 44, 45) | 4.8 (3.0) | -0.7 (2.97)
  Day 28 (n= 45, 45) | -9.2 (3.72) | -13.9 (3.72)
  Day 56 (n= 43, 44) | 1.4 (4.88) | -0.9 (4.82)
  Day 84 (n= 44, 45) | -16.6 (4.71) | -12.1 (4.65)
  Day 126 (n= 45, 45) | 1.6 (4.84) | -1.1 (4.84)
  End of Study (n = 45, 45) | -2.2 (7.25) | 4.9 (7.25)

14. Secondary Outcome: Insulin Resistance as Measured by the Homeostatic Model Assessment (HOMA-IR)
Description: Insulin Resistance is measured via the Homeostatic Model Assessment (HOMA-IR) using a computer to model insulin sensitivity. Insulin Sensitivity (HOMA-%S), where 100% is normal, is the reciprocal of insulin resistance (100/S%). HOMA IR = [fasting insulin (μU/mL)] x [fasting plasma glucose (mmol/L)] / 22.5 where fasting insulin (or glucose) was defined as the arithmetic mean of the -15, -10 and 0 min pre-glucose load values. Analysis of covariance with treatment as a fixed effect and baseline as the covariate was performed on log transformed data.
Time Frame: Baseline, Day 28, Day 84
Population: as for outcome 1
Measure: Geometric Mean (Standard Error); unit: units on a scale
Arm/Group | Cohort 2: Canakinumab Infusion 10 mg/kg | Cohort 2: Placebo to Canakinumab 10 mg/kg | Cohort 3: Canakinumab Infusion 0.1 mg/kg | Cohort 3: Canakinumab Infusion 0.3 mg/kg | Cohort 3: Canakinumab Infusion 1.5 mg/kg | Pooled (Cohort 3 and 4): Placebo Infusion | Cohort 4: Canakinumab Injection 0.03 mg/kg
Number analyzed (Participants) | 45 | 45 | 25 | 24 | 23 | 34 | 20
units on a scale
  Day 28 (n= 44, 45, 24, 24, 22, 33, 20) | 3.30 (0.059) | 3.74 (0.058) | 4.03 (0.092) | 3.34 (0.091) | 3.31 (0.095) | 3.25 (0.078) | 3.31 (0.101)
  Day 84 (n= 44, 45, 24, 24, 23, 33, 20) | 3.37 (0.054) | 3.62 (0.053) | 3.87 (0.103) | 3.43 (0.101) | 4.09 (0.103) | 3.06 (0.087) | 2.94 (0.113)

15. Secondary Outcome: β-cell Function as Measured by the Homeostatic Model Assessment (HOMA-β )
Description: β cell function is measured by the Homeostatic Model Assessment(HOMA-β) using a computer to model β cell function and insulin sensitivity . β cell function is related to Insulin Sensitivity (HOMA-%S) and is the reciprocal of insulin resistance (100/S%). HOMA β = [20 x fasting insulin (μU/mL)] / [fasting plasma glucose (mmol/L) - 3.5] where fasting insulin (or glucose) was defined as the arithmetic mean of the -15, -10 and 0 min pre-glucose load values. Analysis of covariance with treatment as a fixed effect and baseline as the covariate was performed on log transformed data.
Time Frame: Baseline, Day 28, Day 84
Population: as for outcome 1
Measure: Geometric Mean (Standard Error); unit: percent β-cell Function
Groups:
- Pooled (Cohort 3 and 4) : Placebo Infusion: Pooled placebo from cohort 3 and 4. Single dose IV infusion of Placebo
- Cohort 4: Anakinumab Injection 0.03 mg/kg: Single dose IV injection of Canakinumab 0.03 mg/kg
Arm/Group | Cohort 2: Canakinumab Infusion 10 mg/kg | Cohort 2: Placebo to Canakinumab 10 mg/kg | Cohort 3: Canakinumab Infusion 0.1 mg/kg | Cohort 3: Canakinumab Infusion 0.3 mg/kg | Cohort 3: Canakinumab Infusion 1.5 mg/kg | Pooled (Cohort 3 and 4) : Placebo Infusion | Cohort 4: Anakinumab Injection 0.03 mg/kg
Number analyzed (Participants) | 45 | 45 | 25 | 24 | 23 | 34 | 20
percent β-cell Function
  Day 28 (n= 44, 45, 24, 24, 22, 33, 20) | 40.2 (0.05) | 35.9 (0.05) | 38.1 (0.10) | 38.2 (0.10) | 42.0 (0.11) | 37.9 (0.09) | 38.3 (0.11)
  Day 84 (n= 44, 45, 24, 24, 23, 33, 20) | 35.6 (0.06) | 34.3 (0.06) | 34.6 (0.10) | 37.6 (0.10) | 43.3 (0.10) | 37.2 (0.09) | 33.7 (0.11)

16. Secondary Outcome: Number of Participants Reporting Death, Serious Adverse Events (SAEs), Adverse Events (AE) Above 5% Frequency
Description: An adverse event is any unwanted event, whether related to study drug or not occurring during the study period. A Serious Adverse Event (SAE) is an event resulting in death, requiring or prolonging hospitalization, a congenital anomaly or other important medical event. AEs and SAEs were recorded at each visit.
Time Frame: Baseline to End of Study (56[+/-2] and 168 [+/- 5] days after dosing for Cohort 1 and Cohorts 2-4, respectively)
Population: All randomized participants who received study medication were included in the Safety Analysis
Measure: Number; unit: Participants
Arm/Group | Cohort 1: Canakinumab Infusion 0.3 mg/kg | Cohort 1: Placebo to Canakinumab 0.3 mg/kg | Cohort 2: Canakinumab Infusion 10 mg/kg | Cohort 2: Placebo to Canakinumab 10 mg/kg | Cohort 3: Canakinumab Infusion 0.1 mg/kg | Cohort 3: Canakinumab Infusion 0.3 mg/kg | Cohort 3 : Canakinumab Infusion 1.5 mg/kg | Cohort 3: Placebo Infusion | Cohort 4 : Canakinumab Injection 0.03 mg/kg | Cohort 4: Placebo to Canakinumab 0.03 mg/kg
Number analyzed (Participants) | 10 | 5 | 45 | 45 | 25 | 24 | 23 | 24 | 20 | 10
Participants
  Serious Adverse Events | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
  Adverse Events Above 5 % Frequency | 1 | 2 | 9 | 6 | 4 | 4 | 2 | 6 | 10 | 2
  Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Cohort 1: Canakinumab Infusion 0.3 mg/kg | Cohort 1: Placebo to Canakinumab 0.3 mg/kg | Cohort 2: Canakinumab Infusion 10 mg/kg | Cohort 2: Placebo to Canakinumab 10 mg/kg | Cohort 3: Canakinumab Infusion 0.1 mg/kg | Cohort 3: Canakinumab Infusion 0.3 mg/kg | Cohort 3 : Canakinumab Infusion 1.5 mg/kg | Cohort 3: Placebo Infusion | Cohort 4 : Canakinumab Injection 0.03 mg/kg | Cohort 4: Placebo to Canakinumab 0.03 mg/kg
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/5 | 1/45 | 2/45 | 0/25 | 0/24 | 0/23 | 0/24 | 0/20 | 0/10
Other Adverse Events (participants affected / at risk) | 1/10 | 2/5 | 9/45 | 6/45 | 4/25 | 4/24 | 2/23 | 6/24 | 10/20 | 2/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Canakinumab Infusion 0.3 mg/kg (N=10) | Cohort 1: Placebo to Canakinumab 0.3 mg/kg (N=5) | Cohort 2: Canakinumab Infusion 10 mg/kg (N=45) | Cohort 2: Placebo to Canakinumab 10 mg/kg (N=45) | Cohort 3: Canakinumab Infusion 0.1 mg/kg (N=25) | Cohort 3: Canakinumab Infusion 0.3 mg/kg (N=24) | Cohort 3 : Canakinumab Infusion 1.5 mg/kg (N=23) | Cohort 3: Placebo Infusion (N=24) | Cohort 4 : Canakinumab Injection 0.03 mg/kg (N=20) | Cohort 4: Placebo to Canakinumab 0.03 mg/kg (N=10)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal polyp (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Canakinumab Infusion 0.3 mg/kg (N=10) | Cohort 1: Placebo to Canakinumab 0.3 mg/kg (N=5) | Cohort 2: Canakinumab Infusion 10 mg/kg (N=45) | Cohort 2: Placebo to Canakinumab 10 mg/kg (N=45) | Cohort 3: Canakinumab Infusion 0.1 mg/kg (N=25) | Cohort 3: Canakinumab Infusion 0.3 mg/kg (N=24) | Cohort 3 : Canakinumab Infusion 1.5 mg/kg (N=23) | Cohort 3: Placebo Infusion (N=24) | Cohort 4 : Canakinumab Injection 0.03 mg/kg (N=20) | Cohort 4: Placebo to Canakinumab 0.03 mg/kg (N=10)
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ocular hyperaemia (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 7 | 2 | 4 | 2 | 1 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 3 | 2 | 0 | 1 | 0 | 2 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary, however, Novartis does not prohibit any investigator from publishing. Any publications from a single site are postponed until the publication of the pooled data ( i.e., data from all sites ) in the clinical trial.